CLINICAL TRIAL: NCT03589196
Title: Ejaculation Preserving Photoselective Vaporization Versus Plasma Kinetic Vaporization Versus Transurethral Resection Of The Prostate For Management Of Benign Prostatic Enlargement: An Objective Evaluation Through a Prospective Randomized Trial
Brief Title: Ejaculation Preserving Photoselective Vaporization Versus Plasma Kinetic Vaporization Versus Transurethral Resection Of The Prostate: A RCT
Acronym: EPPROSTATECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS/18.02.30
Record Dates: First submitted 2018-05-20; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-03

CONDITIONS: Ejaculation Abnormal; BPH With Urinary Obstruction; Prostatic Hyperplasia; Prostate Disease; Prostate Obstruction
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Photoselective Vaporization (Active Comparator)
  Interventions: Procedure: Ejaculation Preserving Photoselective Vaporization
- Plasma Kinetic Vaporization (Active Comparator)
  Interventions: Procedure: Ejaculation Preserving Plasma Kinetic Vaporization
- Transurethral Resection Of The Prostate (Active Comparator)
  Interventions: Procedure: Ejaculation Preserving Transurethral Resection Of The Prostate

INTERVENTIONS:
Procedure: Ejaculation Preserving Photoselective Vaporization — Ejaculation Preserving Photoselective Vaporization
  Arms: Photoselective Vaporization
Procedure: Ejaculation Preserving Plasma Kinetic Vaporization — Ejaculation Preserving Plasma Kinetic Vaporization
  Arms: Plasma Kinetic Vaporization
Procedure: Ejaculation Preserving Transurethral Resection Of The Prostate — Ejaculation Preserving Transurethral Resection Of The Prostate
  Arms: Transurethral Resection Of The Prostate

SUMMARY:
To Evaluate and compare the outcome and coast of ejaculation sparing management of BPH using 3 different techniques: PVP, PKVP and TURP. Ejaculation sparing TURP group is considered the standard control group. Evaluation will be carried out through a prospective randomized powered trial

ELIGIBILITY:
Inclusion Criteria:

* 1. Age >50 years 2. Prostate volume (measured by TRUS): 30-80 gm 3. International prostate symptom score (IPSS )>15 and quality of life score (QOL)< 3.

  4. Maximum flow rate of uroflometry <10 ml/second 5. Patients with active sexual life (or interested) and having the ability to ejaculate and desire to preserve ejaculation.

  6. Failure or intolerance to medical treatment, recurrent urinary infection, urine retention, significant hematuria or deterioration of the upper urinary tract function secondary to BOO.

Exclusion Criteria:

1. Bleeding disorders and patients on anticoagulant treatment
2. Histologically proved cancer prostate
3. Neurogenic voiding dysfunction
4. Lower urinary tract malignancy
5. Preoperative ejaculation or sexual dysfunction
6. Presence of stricture urethra
7. Unfit for spinal anathesia -

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2018-03-10 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
estimate and compare the ejaculation preservation effect of the 3 techniques (PKVP, PVP and TURP). | 1 years
  assessed by Male Sexual Health Questionnaire (MSHQ)

SECONDARY OUTCOMES:
change in flow rate | 1 years
  measured by uroflowmetery in ml/sec
postoperative complication | 1 year
  measured by Clavien-Dindo Classification scale
change in patients' symptoms. | 1 year
  measured by International Prostate Symptom Score (I-PSS)

CONTACTS AND LOCATIONS:
Locations (1):
- Urology & Nephrology Center, Al Mansurah, Egypt